CLINICAL TRIAL: NCT00372281
Title: Comparison of Cliavist Enhancement in Infectious and Degenerative Diseases of the Spine
Brief Title: Cliavist in Infectious and Degenerative Diseases of the Spine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Direction de la Recherche Clinique et de l'Innovation - Hôpitaux Universitaires de Strasbourg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3780
Record Dates: First submitted 2006-09-04; First posted 2006-09-06 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Spine Infection
Keywords: MRI, CLIAVIST, MACROPHAGE, INFECTION, SPINE
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cliavist (Experimental)
  Interventions: Drug: Cliavist

INTERVENTIONS:
Drug: Cliavist — Injection of 0,9 mL (weight < 60kg) or 1,4 mL (weight > 60kg) of Cliavist (ferucarbotran) by direct intraveinous way, 48 h following the MRI done with gadolinium.

SUMMARY:
USPIO contrast enhancement results from intracellular trapping of the iron particles in reactive cells, especially macrophages. 17FDG-PET studies have demonstrated that macrophages are present in spine infectious diseases but are absent in spine degenerative diseases. The aim of this work is to compare the enhancement induced by CLIAVIST in both diseases. The absence of macrophages in degenerative lesions should help to differentiate them from infectious lesions, who should present contrast enhancement in relation to the presence of macrophages.

ELIGIBILITY:
Inclusion Criteria:

* spine infection or spine degenerative disease
* patient agreement obtained

Exclusion Criteria:

* pregnancy
* MRI contra-indications
* cliavist contra-indication
* dextran allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
First MRI: performed immediately after gadolinium administration | immediately after gadolinium administration
Second MRI: performed 24 hours after cliavist administration | 24 hours after cliavist administration

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Dietemann, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (4):
- France (4):
  - Service de Neuroradiologie - Hôpital Central, Nancy
  - Nouvel Hôpital Civil, Strasbourg
  - Service de Radiologie 2 - Hôpital de Hautepierre, Strasbourg
  - Service de Rhumatologie - Hôpital de Hautepierre, Strasbourg